CLINICAL TRIAL: NCT04258735
Title: Genetic Characteristics of Metastatic Breast Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Young-Hyuck Im, Professor, Samsung Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019-05-157
Record Dates: First submitted 2019-07-23; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metastatic breast cancer cohort (Other): Metastatic breast cancer with genetic tests including WES, RNASeq, ctDNA and exosome
  Interventions: Diagnostic Test: Genomic analysis

INTERVENTIONS:
Diagnostic Test: Genomic analysis — WES, RNASeq, ctDNA, Exosome

SUMMARY:
Genomic analysis for metastatic breast cancer(MBC) patients

* Participant (Inclusion criteria)

  1. Patients who diagnosed metastatic/stage IV breast cancer
  2. Patients who were not received treatment for metastatic breast cancer on palliative setting
* Process

  (1) Tissue/ Blood sample
* At diagnosis, MBC tissue / blood sample (20cc) will be obtained.
* At disease progression after 1st line treatment for MBC, blood sample (20cc) will be obtained (tissue; optional)

  (2) WES, RNASeq, ctDNA, Exosome
* We will analyze genomic characteritics using WES, RNASeq, ctDNA, Exosome.

ELIGIBILITY:
Inclusion Criteria:

* Patients who diagnosed ad metastatic breast cancer
* Patients who were not received treatment on palliative setting

Exclusion Criteria:

* Patients who did not agree this study
* Patients who did not have any pathologic specimen at MBC diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-07-17 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Genomic profiling of MBC patients | 60 months
  Gemetic alteration frequency, the association between genetic alteration and survival

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided